CLINICAL TRIAL: NCT01697553
Title: Home-Based Technologies Coupled to Teleassistance Service: Efficacy for Preventing Falls at Home in Frail Elderly Population Losing Autonomy
Brief Title: Home-Based Technologies Coupled to Teleassistance Service in the Elderly
Acronym: DOMOLIM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: I11 001
Record Dates: First submitted 2012-09-28; First posted 2012-10-02 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Disablement in the Elderly
MeSH Terms: interventions — Home Care Services

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Home automation pack coupled to teleassistance service (Experimental)
  Interventions: Other: home automation pack coupled to teleassistance service
- Home without automation pack coupled to teleassistance service (Active Comparator)
  Interventions: Other: Home without automation pack coupled to teleassistance service

INTERVENTIONS:
Other: home automation pack coupled to teleassistance service
  Arms: Home automation pack coupled to teleassistance service
Other: Home without automation pack coupled to teleassistance service
  Arms: Home without automation pack coupled to teleassistance service

SUMMARY:
The growth of the elderly population is associated with the autonomy failure and the increase of dependence problems. Fall incidents are the third cause of chronic disablement in older persons and are one of the major risk factors for entering in dependence.

The recent progress in home technologies and medical care are opportunities to search how to apply these tools to reduce and prevent falling at home.

The purpose of this study is to evaluate the cost effectiveness of simple home automation pack coupled to teleassistance service for preventing home falls in frail elderly population.

1200 patients will be enrolled and randmosied within two arms:

* home with automation pack coupled to teleassistance service
* home without this technology

DETAILED DESCRIPTION:
This study is one of the first European randomized studies using the criteria MAST (Model for Assessment of Telemedicine) for medico-economic evaluation of technology solutions for the prevention and care in the elderly. The medico-economic evaluation of the overall contribution of home automation kit associated with telecare will be conducted in accordance with the recommendations of the research program Renewing Health FP7 the European Union. This program has developed an analytical model common to all evaluations of telemedicine applications that have an impact on health.

. The home-based technology in this study will be a simple home automation pack coupled to teleassistance service. The automation pack will include: a remote intercom, an electronic bracelet or pendentive, a pull shower in the bathroom, a light path, a smoke detector and a gas detector in the kitchen. The central hotline will provide telephone support at all times.

Intercom is a remote transmitter which enables the platform to provide remote assistance with the elderly at home.

Each person will have electronic bracelet or pendentive with a medallion which will be provided with the dialer. It is a system that allows remote assistance to the elderly by pressing the central medallion of the device to request assistance or report a dangerous situation (risk of falling, or fall) to the platform of teleassistance.

The bathroom alarm zipper is a device installed in the shower that allows subjects to use it when at risk of falling or fall detection. The shower is a high risk of fall for the elderly due to movements very often results in an imbalance of seniors already weakened by aging.

The light path is a 1.5 m device installed near the bed and turns automatically on when the person sets foot on the ground. It can provide adapted visibility by showing the right path and improving consciousness.

The smoke and gas detector are devices installed on the ceiling of the kitchen. They allow respectively detecting abnormally high rates of smoke or a gas leak in the house or apartment.

The teleassistance platform is a central technical hotline located in Creuse area. It is functional at any time. All electronic devices are connected to the plant. An alert is signaled by an alarm, involving an immediate phone call to the resident of the house to assess the situation. The resulting actions taken are either reassuring the person, giving directions to the person or sending a message to aid in the event ascertained or suspected.

A monthly questionnary should be filled by patients.

Primary outcome:

The main judgment criterion will be the cumulated incidence of home falls requiring emergency admission.

Secondary outcomes:

1. Changes score ISO profile resource according to SMAF scale,
2. Proportion of participants with regular physical activity
3. Effect on admissions in institutions (nursing homes or senior residential care)
4. Time before management of stroke and the length of stay in rehabilitation unit.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 65 or over
* Living at least for 1 year in the department of Creuse
* Frail elderly or pre-frail according to the criteria of Fried
* Patient with autonomy enough to get out of bed
* Having a cognitive level acceptable (MMS ≥ 10)
* Place of life arranged and adapted to the installation of the DSTA
* Consentbsigned by the patient and / or its trusted person or his legal representative
* Affiliation or beneficiary of a social security system

Exclusion Criteria:

* Patient under guardianship or protection of justice
* patient home already equiped with automation pack different from theone of the experiment
* People who can not read or write
* Diseases involving life-threatening in the short term (<1 year)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2012-10; Primary Completion 2015-10 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
incidence of home falls requiring emergency admission | at 12 months
  The cumulated incidence of home falls requiring emergency admission.

SECONDARY OUTCOMES:
Changes score ISO profile resource according to SMAF scale | at 12 months
Proportion of participants with regular physical activity | at 12 months
Effect on admissions in institutions (nursing homes or senior residential care) | at 12 months
Time before management of stroke and the length of stay in rehabilitation unit | at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Thierry DANTOINE, MD, Study Chair — CHU Limoges
Locations (4):
- France (4):
  - CH Aubusson, Aubusson
  - CH Bourganeuf, Bourganeuf
  - CH de Gueret, Guéret
  - CHU Limoges, Limoges